CLINICAL TRIAL: NCT07390331
Title: A Theory-Informed, Brief Patient Activation and Motivational Interviewing Approach to Implementing Depression Treatment in Cardiac Patients: A Quality Improvement Initiative
Brief Title: A Patient Activation Approach to Implementing Depression Treatment in Cardiac Patients
Acronym: iHeart_2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nathalie Moise, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAV9954; P30AG064198 (NIH)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Depression and CVD
Keywords: patient activation; depression treatment uptake; depression treatment optimization
MeSH Terms: conditions — Depression; Cardiovascular Diseases; Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening alone (No Intervention): As part of a Quality Improvement Initiative, navigators and clinical staff call patients to screen patients for depression using the Patient Health Questionnaire (PHQ)-2 followed by the PHQ-9 in advance of scheduled office visits with cardiologists or primary care clinicians and enter results into Epic for providers to view during their visits and refer and manage depression at their discretion. Patients will receive the clinic's mental health informational resource.
- Screening plus iHeart DepCare tool and Motivational Interviewing (Active Comparator): As part of a Quality Improvement Initiative, navigators and clinical staff call patients to screen patients for depression using the Patient Health Questionnaire (PHQ)-2 followed by the PHQ-9 in advance of scheduled office visits with cardiologists or primary care clinicians and enter results into Epic for providers to view during their visits and refer and manage depression at their discretion.
  Eligible patients who screen positive for depression (PHQ-9 ≥8) are administered the Heart DepCare tool along with motivational, technical and navigational support per patient preference. Clinical and mental health providers are sent the patient's treatment preferences via EPIC.
  Interventions: Behavioral: iHeart Depcare tool

INTERVENTIONS:
Behavioral: iHeart Depcare tool — The iHeart DepCare tool is an electronic patient activation and psychoeducation tool (available in English and Spanish) designed to bridge depression screening with treatment. The tool includes: 1) a description of depressive symptoms; 2) a checklist of behavioral risk factors; 3) an animation of a CVD patient going through the process of symptom recognition, help seeking, and treatment completion following a CVD event; 4) psychoeducation videos; 5) depression treatment selection support (adapted to include behavioral risk factor preferences); and 6) additional cardiac resources the patient can reference. Patients may receive brief motivational interviewing as well as technical/navigational support per patient preference to reinforce learning. Patient treatment preferences are sent via EPIC to the mental health and treating providers.
  Arms: Screening plus iHeart DepCare tool and Motivational Interviewing

SUMMARY:
This study, which is being conducted as part of a Quality Improvement (QI) Initiative at Columbia University Irving Medical Center, will test whether delivering the iHeart DepCare tool increases real world reach and adoption of depression treatment among CHD patients. As part of the QI Initiative, Clinic Navigators will administer and record (in EPIC) depression screening in advance of primary care and cardiology appointments. Eligible patients with elevated depressive symptoms will be randomized to receive usual care vs. the iHeart DepCare tool in conjunction with brief motivational, technical and navigation support per patient preference.

Aim 1: To test the effect of iHeart DepCare on depression treatment optimization (primary outcome) among coronary heart disease patients with elevated depressive symptoms.

Aim 2: To explore the effect of iHeart DepCare on implementation outcomes, including provider referrals, among coronary heart disease patients with elevated depressive symptoms.

DETAILED DESCRIPTION:
Depression is common in patients with coronary heart disease (CHD) and associated with increased cardiac morbidity and mortality. Evidence-based mental health treatment improves depressive symptoms and quality of life, yet few CHD patients engage in treatment. The investigator previously tested the efficacy of an implementation strategy centered around a patient activation and psychoeducation tool (iHeart DepCare) for improving depressive symptoms and uptake of depression treatment in CHD patients. The research now expands to test the real-world effectiveness of the iHeart DepCare tool in cardiology and primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* PHQ9 or PHQ8 score >=8
* History of coronary heart disease per EHR search for ICD-9 codes of 410-414 and ICD-10 codes: I20, I21, I22, I23, I24, I25.
* Appointment with a primary care provider (PCP) or cardiologist in an integrated care setting in NYP/Columbia (e.g., does not include procedure or lab-only visits)
* Has a PCP at NYP/Columbia active on the NYP/Columbia EHR

Exclusion Criteria:

* Not English or Spanish speaking
* History of severe mental illness (bipolar disorder, schizophrenia, chronic/recurrent depression, history of suicide attempt or self-inflicted injuries)
* Dementia
* Had an integrated mental health visit in the last 3 months as indicated in the EHR
* Enrollment in the post-implementation period of IRB# AAAR9175

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of eligible patients who initiate or intensify depression treatment | Up to 6 months
  This is designed to measure depression treatment reach, which is defined as the percentage of eligible patients who initiate or intensify depression treatment within 6 months of the index visit, as indicated by ≥1 pharmacy fill data of a new or changed antidepressant and/or a new visit with a mental health provider (e.g., psychologist, psychiatrist, behavioral health provider like social workers) and/or primary care provider with a visit diagnosis of depression and/or an exercise program (e.g., cardiac rehabilitation), which will be assessed through chart extraction and tallied.

SECONDARY OUTCOMES:
Percentage of patients in whom their clinician referred to mental health treatment | Baseline
  This is designed to measure treatment adoption, which is defined as the percentage of patients in whom their clinician referred to mental health treatment (e.g., collaborative care, psychotherapy, psychiatry, cardiac rehab) and/or prescribed/changed antidepressants and/or psychological/supportive counseling at the index visit, which will be assessed through chart extraction and tallied.
Mean adherence to cardiac medications | Approximately between 3 to 9 months from baseline
  Mean adherence will be assessed as the mean proportion of days covered (PDC) for key cardiovascular disease medications (i.e., statin, antihypertensives) based on fill dates in the 3-9 months after the index visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Moise, MD, MS, FAHA, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States